CLINICAL TRIAL: NCT00180336
Title: CONTAK RENEWAL 4 AVT Field Following
Brief Title: Safety and Efficacy Study of RENEWAL 4 AVT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0004
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Heart Failure; Tachycardia; Atrial Fibrillation; Atrial Flutter; Ventricular Fibrillation
Keywords: Heart Failure; Tachycardia; Atrial Fibrillation; Atrial Flutter; Ventricular Fibrillation
MeSH Terms: conditions — Heart Failure; Tachycardia; Atrial Fibrillation; Atrial Flutter; Ventricular Fibrillation

INTERVENTIONS:
Device: CRT-D

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the CONTAK RENEWAL 4 AVT device.

DETAILED DESCRIPTION:
This is a prospective, two-arm, non-randomized, multi-center European field following, designed to demonstrate the safety and effectiveness of the CONTAK RENEWAL 4 AVT device in humans.

ELIGIBILITY:
Inclusion Criteria:

* Indications for the device
* Availability for follow-up at an approved Field Following center, at the protocol defined intervals
* Willing and capable of undergoing a device implant and participating in all testing associated with this clinical investigation
* Prescribed to stable optimal pharmacologic therapy for HF
* Age 18 or above, or of legal age to give informed consent specific to national law
* Able to provide documented evidence of one or more episodes of AF/AT within 12 months of implantation NOTE: Guidant recommends anticoagulation therapy per physician discretion.

Exclusion Criteria:

* Right bundle branch block morphology
* Life expectancy of less than six months due to other medical conditions
* Expectation of a heart transplant during the period of the study
* Patients with or who are likely to receive a mechanical tricuspid valve during the course of the study
* Have a preexisting unipolar pacemaker that will not be explanted/abandoned
* Have an atrial tachyarrhythmia that is permanent (i.e., does not terminate spontaneously and cannot be terminated with medical intervention) within 180 days prior to enrollment
* Have a known hypersensitivity to dexamethasone acetate
* Enrolled in any other study, including drug investigation
* Women that are pregnant or planning to become pregnant
* A Cerebral Vascular Event/ Transient Ischemic Attack within 12 months of implantation
* During the four weeks prior to implantation, a patient experiences an episode of AF >= 48 hours in duration and was not anticoagulated for at an adequate therapeutic level (INR >= 2.0) for the 4 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170
Dates: Start 2004-07

PRIMARY OUTCOMES:
System Complication-Free Rate at 6 months
Effectiveness of LV Only/LV Offset at 6 months

SECONDARY OUTCOMES:
LVESD at 6 months
Six-minute walk at 6 months
NYHA at 6 months
QOL at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sperzel, MD, Principal Investigator — Kerckhoff Klinik Bad Nauheim (Germany)
Locations (1):
- Kerckhof Klinik, Bad Nauheim, Germany